CLINICAL TRIAL: NCT00981292
Title: Cerebral Blood Flow, Cerebro-electrical Activity and Behavioural Effects of Epigallocatechin Gallate (EGCG) Administration in Healthy, Young Adults
Brief Title: Effects of Epigallocatechin Gallate (EGCG) in Healthy, Young Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Crystal Haskell, Research Fellow, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 24Z1
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-03

CONDITIONS: Cognitive Function; Mood
Keywords: Epigallocatechin Gallate; cerebral blood flow; Near Infrared spectroscopy; Electroencephalography; cognitive function; mood; cerebro-electrical activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 135mg EGCG (Active Comparator)
  Interventions: Dietary Supplement: EGCG; Dietary Supplement: Placebo
- 270mg EGCG (Active Comparator)
  Interventions: Dietary Supplement: EGCG; Dietary Supplement: Placebo
- 0mg EGCG (Placebo Comparator)
  Interventions: Dietary Supplement: EGCG; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EGCG — Acute oral administration of capsules containing either: 0mg, 135mg or 270mg. One dosage administered on each of three separate study days.
  Other Names: Teavigo
Dietary Supplement: Placebo — Pharmaceutical grade silica was utilized as placebo

SUMMARY:
Epigallocatechin gallate (EGCG) is the most abundant catechin (sometimes referred to as tea flavonoids) in green tea extract. A review by Nagle et al (2006) identifies that a large amount of research indicates EGCG (amongst other catechins) is responsible for most of the potential health benefits associated with green tea. EGCG is brain permeable (Nakagawa & Miyazawa, 1997), and it is considered to have neuroprotective and neurorescue effects including modulation of cell survival and cell cycle genes (Levites et al 2002).

Although there have been several human studies looking at the bioavailability of EGCG when administered in varying doses, there have been no studies that have specifically investigated the cognitive effects of this catechin in humans. Therefore, the purpose of this study is to assess the cerebral blood flow (using Near Infrared Spectroscopy), cerebro-electrical activity (EEG) and behavioural effects of EGCG. A randomised, double-blind, placebo-controlled, balanced crossover study will assess the effects of 135 mg and 270 mg pure EGCG in 24 healthy, young adults (18-35). Prior to the first active study day participants will attend a screening/training visit where relevant exclusion criteria will be assessed including any food sensitivities. They will also complete a caffeine consumption questionnaire in order to control for potential caffeine withdrawal effects as a result of restrictions of the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* aged 18-35
* either caffeine consumers (consume more than 150mg caffeine per day) or non-consumers (consume less than 44mg caffeine per day).

Exclusion Criteria:

* smoke or consume any tobacco products
* not proficient in English language
* pregnant (or seeking to become pregnant)
* taking recreational, over the counter/prescription medication (including the contraceptive pill), and/or dietary/herbal supplements
* have food allergies or sensitivities
* have history of/current head trauma, learning difficulties , ADHD, migraines or any gastric problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- 135mg EGCG Then 0mg EGCG Then 270mg EGCG; 270mg EGCG Then 135mg EGCG Then 0mg EGCG; 0mg EGCG Then 135mg EGCG Then 270mg EGCG; 135mg EGCG Then 270mg EGCG Then 0mg EGCG; 0mg EGCG Then 270mg EGCG Then 135mg EGCG; 270mg EGCG Then 0mg EGCG Then 135mg EGCG: Those participants who received treatment in this order.
Period: Day 1
Arm/Group | 135mg EGCG Then 0mg EGCG Then 270mg EGCG | 270mg EGCG Then 135mg EGCG Then 0mg EGCG | 0mg EGCG Then 135mg EGCG Then 270mg EGCG | 135mg EGCG Then 270mg EGCG Then 0mg EGCG | 0mg EGCG Then 270mg EGCG Then 135mg EGCG | 270mg EGCG Then 0mg EGCG Then 135mg EGCG
Started | 7 | 4 | 6 | 4 | 4 | 7
Completed | 6 | 4 | 6 | 4 | 4 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 2
Period: Day 2
Arm/Group | 135mg EGCG Then 0mg EGCG Then 270mg EGCG | 270mg EGCG Then 135mg EGCG Then 0mg EGCG | 0mg EGCG Then 135mg EGCG Then 270mg EGCG | 135mg EGCG Then 270mg EGCG Then 0mg EGCG | 0mg EGCG Then 270mg EGCG Then 135mg EGCG | 270mg EGCG Then 0mg EGCG Then 135mg EGCG
Started | 6 | 4 | 6 | 4 | 4 | 5
Completed | 4 | 4 | 6 | 4 | 4 | 5
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0
Period: Day 3
Arm/Group | 135mg EGCG Then 0mg EGCG Then 270mg EGCG | 270mg EGCG Then 135mg EGCG Then 0mg EGCG | 0mg EGCG Then 135mg EGCG Then 270mg EGCG | 135mg EGCG Then 270mg EGCG Then 0mg EGCG | 0mg EGCG Then 270mg EGCG Then 135mg EGCG | 270mg EGCG Then 0mg EGCG Then 135mg EGCG
Started | 4 | 4 | 6 | 4 | 4 | 5
Completed | 4 | 4 | 6 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 135mg EGCG Then 0mg EGCG Then 270mg EGCG | 270mg EGCG Then 135mg EGCG Then 0mg EGCG | 0mg EGCG Then 135mg EGCG Then 270mg EGCG | 135mg EGCG Then 270mg EGCG Then 0mg EGCG | 0mg EGCG Then 270mg EGCG Then 135mg EGCG | 270mg EGCG Then 0mg EGCG Then 135mg EGCG | Total
Number analyzed (Participants) | 7 | 4 | 6 | 4 | 4 | 7 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 6 | 4 | 4 | 7 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22 (4) | 22 (4) | 22 (4) | 22 (4) | 22 (4) | 22 (4) | 22 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 3 | 3 | 2 | 18
  Male | 3 | 1 | 3 | 1 | 1 | 5 | 14
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 4 | 6 | 4 | 4 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Modulation of Levels of Total Haemoglobin
Description: This measure assessed changes in levels of total haemoglobin during the 42 minute post- dose task period. Levels are in μmol/L and represent change from baseline levels.
Time Frame: 42 minutes
Population: If NIRS readings were deemed not too affected by artefacts (usually caused by participants moving the headband in some way) then they were utilized in the analysis.
Measure: Mean (Standard Error); unit: μmol/L
Groups:
- 135mg EGCG: All participants when consumed 135mg EGCG.
- 270mg EGCG: All participants when consumed 270mg EGCG.
- Placebo: All participants when consumed Placebo.
Arm/Group | 135mg EGCG | 270mg EGCG | Placebo
Number analyzed (Participants) | 27 | 27 | 27
μmol/L | -1.4 (0.5) | -1.3 (0.3) | -1.7 (0.3)
Statistical Analysis 1: Comparison: 135mg EGCG; This data was analysed by two-way repeated measures ANOVA (task [epoch] x treatment). In the case of those analyses that showed a significant main effect of treatment or a task/epoch x treatment interaction, planned comparisons of data from each task or epoch were then made between placebo and each of the EGCG treatment groups using t tests calculated with the Mean Squares Error from the ANOVA; Test type: Superiority or Other; p < 0.05, ANOVA — A Bonferroni adjustment was made for multiplicity

2. Secondary Outcome: Number of Participants With Significant Modulation of Cognitive Performance
Description: The cognitive performance of participants was assessed via a range of computerised, mentally demanding, executive function tasks: Serial 3s and 7s subtractions, oddball reaction time task, rapid visual information processing, stroop and simple reaction time.These tasks were completed at baseline and then again 45 minutes after treatment administration. Significant modulation was determined if participants' post dose scores were significantly higher than baseline.
Time Frame: 42 minutes
Population: If participants were deemed to have completed the tasks to the best of their ability then their scores were utilized in the analysis.
Measure: Number; unit: Participants
Groups:
- 135mg: All participants when consumed 135mg EGCG.
Arm/Group | 135mg | 270mg EGCG | Placebo
Number analyzed (Participants) | 27 | 27 | 27
Participants | 0 (0) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: 135mg vs 270mg EGCG vs Placebo; Task performance data were analysed by within subjects ANCOVA (treatment) with pre-treatment performance included as a co-variate for each individual task/measure; Test type: Superiority or Other; p > 0.05, ANCOVA

3. Secondary Outcome: Number of Participants With Significant Modulation of Mood.
Description: Mood was assessed via computerised visual analogue scales at baseline and post- dose time points. Mood scores were calculated as change from baseline. And significant modulation was determined if baseline scores were significantly different to post dose.
Time Frame: 42 minutes
Population: As long as data for all participants was captured for all 3 sessions then that participants data was utilized in the analysis.
Measure: Number; unit: Participants
Arm/Group | 135mg EGCG | 270mg EGCG | Placebo
Number analyzed (Participants) | 27 | 27 | 27
Participants | 0 (0) | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: 135mg EGCG vs 270mg EGCG vs Placebo; Mood data was analysed via student t-test; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | 135mg EGCG Then 0mg EGCG Then 270mg EGCG | 270mg EGCG Then 135mg EGCG Then 0mg EGCG | 0mg EGCG Then 135mg EGCG Then 270mg EGCG | 135mg EGCG Then 270mg EGCG Then 0mg EGCG | 0mg EGCG Then 270mg EGCG Then 135mg EGCG | 270mg EGCG Then 0mg EGCG Then 135mg EGCG
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/6 | 0/4 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/6 | 0/4 | 0/4 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No